CLINICAL TRIAL: NCT00857987
Title: Randomized , Placebo-controlled, Clinical Trial of Efficacy and Safety Evaluation of Guaifenesin, Doxylamine Succinate and Hydrochloride Etafedrine Syrup in Improving the Signs and Symptoms of Infections of Way Upper (URI)
Brief Title: Effectiveness and Safety of the of Guaifenesin, Doxylamine Succinate and Hydrochloride Etafedrine Syrup in Improvement of Symptoms Resulting From Acute Respiratory Infections.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GADEMS0109; GADEMS0109
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Upper Airway Infections
Keywords: IRA, Guaifenesin, Etaphedrine, Doxilamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Guaifenesin, doxylamine succinate and hydrochloride etafedrine syrup
  Interventions: Drug: EMS Expectorant
- 2 (Placebo Comparator): Vehicle
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: EMS Expectorant — Guaifenesin - 100mg, Etafedrine hydrochloride 20mg, Succinate doxilamine 6mg.
  Arms: 1
Other: Placebo — Vehicle
  Arms: 2

SUMMARY:
Evaluate the improvement of the common cold with the use of medication

DETAILED DESCRIPTION:
Patients with signs and symptoms of URI will be forwarded to the Research Center for a screening in which the researchers will select those meet the inclusion criteria. This visit will be informed of the objectives study, methodology, risks and benefits, the right of patients to give up research, the confidentiality of data and other details that provide the the patients to consider their participation basement viable or not. All aspects relevant to the consideration of the patient on their participation will described in the Informed Consent, which will be read and signed before any procedure. The patients included are randomized, open treatment immediately and will be sent to perform a radiological examination (Rx - sinus of the face). This examination used to detect other clinical pictures than URI. After 24 hours (visit 02), the patient will return for the assessment and clinical questions about their symptoms, which provide the scores of efficacy of the product. This visit will review the radiological examination, and on the finding that infection of sinuses without symptoms, the patient will excluded because of antibiotic use will begin. In return for three days (visit 03), patients will again evaluated in relation to their clinical status. On this visit, the doctor may take the following behaviors:

* Patients who have no clinical symptoms get high.
* Patients who have not improved, take a dose of medicine increased.
* The worsening of the present that, due to infections bacterial or other clinical pictures, will be excluded and referred to a general practitioner employed by the sponsor. In return for seven days, patients should return the products and again participate in a clinical consultation, in which researchers may take the following behaviors:
* Patients who have no clinical symptoms get high.
* Patients who have not improved or have worsened will be exempted from study and referred to the general practitioner hired by the sponsor is repeated for the diagnosis and establish a new treatment. Will be allowed the use of rescue medications such as paracetamol or sodium dipyrone, justified by the existence of the placebo group and those products do not interfere in the results evaluated, it was a pain and antipyretics.

ELIGIBILITY:
Inclusion Criteria:

* Patients who take part in the study, agreeing with the terms proposed in FICT;
* Patients aged 12 years or above of any ethnicity, class or social group;
* Patients of both sexes;
* Patients with good mental health;
* Patient with acute respiratory disease of the upper airways of viral etiology (URI);
* Patient with the early signs and symptoms of URI with minimum time of failure greater than 48 hours.

Exclusion Criteria:

* Patients treated with antibiotics or predict the use of antibiotics for other clinical condition;
* Presence of bacterial tables of the upper airways and lungs (bacterial sinusitis, pneumonia, etc.).
* Patient with cystic fibrosis;
* Primary or metastatic cancer to the lung;
* Presence of respiratory tables with more than 14 days in duration;
* Treatment with immunosuppressive drugs;
* Presence of any medical or psychological condition that, at the discretion of the investigator, should prevent the patient from the study;
* History of abuse of alcohol or drugs;
* Participation in clinical trials in the six months preceding the study;
* Patients with severe pulmonary diseases, which require multi-drug treatment;
* Presence of other concomitant pulmonary diseases;
* Pregnancy and lactation;
* History of hypersensitivity to drugs of the same pharmacological classes of substances under investigation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
- Decrease in nasal secretion - Decrease in sneezing - Reduction of edema of the nasal mucosa - Decreased frequency of cough - Decrease the frequency of dyspnea - Reduction of nasal obstruction | Screening (Day 0); Return to 1 day; Return to 3 days (+/-1); Return of 7 days (+ / -2)

SECONDARY OUTCOMES:
Will be assessed for safety by the incidence of adverse reactions | Screening (Day 0); Return to 1 day; Return to 3 days (+/-1); Return of 7 days (+ / -2)

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clinica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil